CLINICAL TRIAL: NCT04532034
Title: Facilitating Emerging Adults Engagement in Evidenced-Based Treatment for Early Psychosis Through Peer-Delivered Decision Support
Brief Title: Facilitating Engagement in Evidence-Based Treatment for Early Psychosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 261047; K08MH116101 (NIH)
Record Dates: First submitted 2020-07-21; First posted 2020-08-31 (Actual); Results first posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-03

CONDITIONS: Psychotic Disorders
Keywords: Decision Support Techniques, Young Adult
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Peer-Delivered Decision Support Intervention (Experimental)
  Interventions: Behavioral: Peer-Delivered Decision Support Intervention

INTERVENTIONS:
Behavioral: Peer-Delivered Decision Support Intervention — An intervention provided by a trained peer interventionist to facilitate treatment decision making among emerging adults with early psychosis. Specific components of this intervention may include facilitating access to information, clarifying values, helping a person obtain the needed support to make a decision, and screening for implementation barriers. Due to having lived experience of a mental health condition, the peer interventionist will also be able to provide unique types of information and support within the coaching process.

SUMMARY:
The purpose of this mixed methods study is to evaluate a peer-delivered decision support intervention with emerging adults newly enrolled in an early intervention program, also known as coordinated specialty care (CSC). It is hypothesized that participants will experience a reduction in decision-making needs after participating in the intervention, and that study and intervention procedures will demonstrate feasibility and acceptability.

DETAILED DESCRIPTION:
The overarching goal of this study is to pilot test a peer-delivered decision support intervention (in the form of decision coaching) that is designed to enhance emerging adults' treatment decision-making and service engagement after enrollment in a coordinated specialty care (CSC) program. Based on an experimental therapeutics approach, this mixed methods pilot trial will assess feasibility, acceptability, and the intervention's potential impact on key decision-making needs (i.e., decision-making targets). We will track feasibility data related to study and intervention procedures, and collect acceptability and outcome data from 20 emerging adults who will participate in the intervention after enrollment in the CSC program. Quantitative analysis related to decision-making targets will provide preliminary evidence regarding whether the intervention impacts these targets, while qualitative analysis will explain how it may do so. Merged results from these two sets of data will inform intervention refinement by providing a nuanced understanding of the intervention's potential to engage decision-making targets from the perspective of emerging adults.

ELIGIBILITY:
Inclusion Criteria:

* 18-30 years of age
* Experiencing early psychosis,defined as psychosis lasting 18 months or less between the time when threshold symptom criteria were reached (as determined by the admitting CSC program assessor) and the date of CSC program enrollment
* Able to speak/understand English
* Able to provide informed consent as assessed by research staff
* Enrolled in the CSC program for any period of time

Exclusion Criteria:

* having a legal guardian
* Diagnosis of dementia, delirium, or intellectual disability as determined by the admitting CSC program psychiatrist

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Thomas, Ph.D., Principal Investigator — Temple University
Locations (3):
- United States (3):
  - Child and Family Focus (On My Way Program), Broomall, Pennsylvania
  - CMSU Behavioral Health & Developmental Services, Danville, Pennsylvania
  - Horizon House, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thomas EC, Lucksted A, Siminoff LA, Hurford I, O'Connell M, Penn DL, Casey I, Smith M, Suarez J, Salzer MS. Case Study Analysis of a Decision Coaching Intervention for Young Adults with Early Psychosis. Community Ment Health J. 2025 Jul;61(5):874-889. doi: 10.1007/s10597-024-01425-w. Epub 2025 Jan 3. PMID 39746883
- [Derived] Thomas EC, Suarez J, Lucksted A, Siminoff LA, Hurford I, Dixon LB, O'Connell M, Penn DL, Salzer MS. Facilitating treatment engagement for early psychosis through peer-delivered decision support: intervention development and protocol for pilot evaluation. Pilot Feasibility Stud. 2021 Oct 24;7(1):189. doi: 10.1186/s40814-021-00927-8. PMID 34689830

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Peer-Delivered Decision Support Intervention
Started | 12
Completed | 6
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | Peer-Delivered Decision Support Intervention
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.42 (2.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Participants self-reported whether they belonged to the following racial/ethnic groups: Asian, African American, White, Hispanic/Latino, and Other. Racial and ethnic groups were non-mutually exclusive.
  Participants
    Asian | 2
    African American | 6
    White | 4
    Hispanic/Latino | 1
    Other | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12
Decisional Conflict Scale [Mean (Standard Deviation); unit: units on a scale] — Total scores on the Decisional Conflict Scale are calculated as: (sum of all items scores / the total number of items) x 25. For this study, 9 items were included. Population: Data was missing from 2 participants on the Decisional Conflict Scale at baseline.
  units on a scale
    number analyzed (Participants) | 10
    (all) | 26.39 (7.55)

OUTCOME MEASURES:

1. Primary Outcome: Change in Decisional Conflict Scale
Description: Change was calculated as the Decisional Conflict Scale value at intervention completion minus the value at baseline. Total scores on the Decisional Conflict Scale are calculated as: (sum of all items scores / the total number of items) x 25. For this study, 9 items were included. Scores on the Decisional Conflict Scale range from 0-100, with higher scores indicating a worse outcome.
Time Frame: Baseline, through intervention completion (up to 3 months)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peer-Delivered Decision Support Intervention
Number analyzed (Participants) | 5
score on a scale | 0.55 (18.68)
Statistical Analysis 1: Comparison: Peer-Delivered Decision Support Intervention; Test type: Other; p = .95, t-test, 2 sided; Mean Difference (Final Values) = .067

ADVERSE EVENTS:
Time Frame: Adverse events were assessed at baseline and follow-up. For participants who completed a follow-up interview, assessment of adverse events pertained to the entire period of participants' participation in the study (approximately 3 months).
Arm/Group | Peer-Delivered Decision Support Intervention
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 1/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Peer-Delivered Decision Support Intervention (N=12)
Urinary Tract Infection (Infections and infestations) | 1
Suicidal ideation (Psychiatric disorders) | 1 — Participant indicated that she experienced suicidal ideation and sought crisis services to manage this experience. She indicated that her suicidal ideation was unrelated to her participation in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-22): https://cdn.clinicaltrials.gov/large-docs/34/NCT04532034/Prot_SAP_000.pdf